CLINICAL TRIAL: NCT00774384
Title: A Phase II, Open Label, Randomised, Single Centre Study To Evaluate The Importance Of Naturally Induced Immune Regulation On The Mucosal Immune Response To Meningococcal Serogroup B Outer Membrane Vesicle (Omv) Vaccine When Administered Intramuscularly To Adults & Adolescents
Brief Title: Regulation of Mucosal Immune Response to Systemic MenB Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Collaborators: University of Bristol (Other); Public Health England (Other Government); Novartis Vaccines (Industry); North Bristol NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SysVac01 - C60P2 PA/2008/2883
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Meningococcal Infections
Keywords: Neisseria meningitidis; Mucosal; Vaccination; Immunity; T cells; T regulatory cells
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Immunisation with NZ MenB OMV vaccine (NZ98/254)
  Interventions: Biological: NZ MenB OMV vaccine (NZ98/254)
- 2 (No Intervention): No vaccine

INTERVENTIONS:
Biological: NZ MenB OMV vaccine (NZ98/254) — 3 doses by intramuscular injection
  Arms: 1

SUMMARY:
Meningitis or septicaemia (blood poisoning) caused by group B meningococcal infection (MenB) is an important cause of death and disability in the UK. Prevention through vaccination therefore remains a key public health priority. Research from national "meningitis" vaccine programmes against MenC, Hib and Streptococcus pneumoniae show us that their success is in part due to their ability to protect both the vaccinated and the unvaccinated, so-called herd immunity. This protection probably occurs by reducing carriage of these meningitis bacteria in the back of the throat (mucosal immunity). How this happens is poorly understood but our research shows that naturally acquired immunity (transient contact between the immune system and the meningococcus in the back of the throat without causing disease) may impact on this process. We believe that to develop a MenB vaccine that is able to cause mucosal immunity and prevent MenB carriage, it is important to understand the interaction between natural immunity and vaccination. In this study we propose to administer MenB vaccine to adults in order to investigate this process. Our findings will provide important insights into Men B immunity, inform the design of novel vaccine strategies and allow the rational testing of new vaccines as they become available.

DETAILED DESCRIPTION:
Meningitis or septicaemia (blood poisoning) caused by group B meningococcal infection (MenB) is an important cause of death and disability in the UK. Our research shows that naturally acquired mucosal immunity (transient contact between the immune system and the meningococcus in the back of the throat without causing disease) may impact on the ability of new Men B vaccines to protect both the vaccinated and the unvaccinated, so called herd immunity. We ask the question, do specialised immune cells called CD25+ regulatory T cells (Treg) operating in the back of the throat explain the failure of immunisation to boost mucosal T cell immunity in teenagers and young adults?

PURPOSE & OBJECTIVES: MenB is the commonest cause of bacterial meningitis in the UK, and is a frequent cause of septicaemia in children and young adults. Death may occur in up to 20% of individuals and long term sequelae are frequent amongst those that survive. In contrast to a highly successful MenC vaccine programme, the burden of MenB disease remains considerable. Prevention through vaccination is therefore a key public health priority in the UK. This project will inform the development of a broadly protective MenB vaccine. We propose to: 1) Determine the nature of the mucosal CD25+ Treg population that regulates MenB immunity. 2) Establish whether naturally induced mucosal CD25+ Treg activity in adults and adolescents modulates the mucosal immune response to systemic MenB OMV vaccination. 3) Investigate the impact of this regulation on mucosal B cell memory

DESIGN: This phase II, open label, randomised, single centre study of a MenB vaccine will utilise cells isolated from human tonsils to measure vaccine-induced T cell immune responses to MenB in adults and adolescents. Comparisons will be made with a control unvaccinated population. RECRUITMENT: Ear, Nose and Throat surgeons will be approached to agree to the participation of their patients in the study. Subjects will be invited by letter to express an interest in the study. Interested individuals will then be contacted by study medics who will provide the appropriate subject information sheet. All study visits and clinical procedures will be undertaken at University Hospitals Bristol NHS Foundation Trust, Bristol. Study clinical personnel will then obtain written informed consent for participation from the subject. No study procedure will be undertaken until written informed consent is given. Following confirmation of inclusion and exclusion criteria, subjects will be enrolled in the study.

RANDOMISATION: On inclusion in the study, subjects will be allocated the next available subject number. Subjects enrolled into the study will be assigned a 5-digit subject number. The first two digits identify the study site. The next three digits identify the subject within the site and will be assigned sequentially, with 001 corresponding to the first subject enrolled. The subject number will determine the treatment group to which the subject is randomised according to a computer-generated block randomisation procedure.

INCLUSION / EXCLUSION: Individuals eligible to be enrolled in this study are male and female subjects. The eligibility of subjects to take part in the study will be assessed by a dedicated Vaccine Study doctor or nurse prior to enrolment.

Inclusion criteria:

* written informed consent and agreement for samples to be sent overseas
* adults and adolescents 16-40 years scheduled to undergo routine tonsillectomy
* in good health at the time of entry into the study as determined by medical history, physical examination and clinical judgment of the investigator
* availability for all the visits scheduled in the study

Exclusion criteria:

* tonsillectomy for allergic conditions
* receipt of or intent to immunize with any vaccination (other than influenza vaccine or post-exposure tetanus vaccination) or investigational agents within 50 days prior to enrolment and throughout the study period
* previous receipt of any MenB vaccine
* chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs (Inhaled and topical steroids will not be allowed.)
* history of confirmed or suspected meningococcal infection or close contact with an individual with culture or PCR proven N. meningitidis serogroup B within the previous 60 days
* pregnancy (or plans to become pregnant during study)* or breast feeding
* not taking or unwilling to take sufficient measures to avoid pregnancy occurring for the duration of the study period**
* any chronic or progressive disease (eg neoplasm, cardiac, respiratory, liver, gastrointestinal, renal, neurological disease, autoimmune disease, blood dyscrasias or diathesis) or history of dependence/abuse of drugs or alcohol • any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* administration of immunoglobulins and/or any blood products in the last year or planned administration during the study period
* history of any anaphylactic shock, asthma, urticaria or any other allergic reaction after previous vaccinations, or known hypersensitivity to any vaccine component
* fever (oral temperature equal to or greater than 38.5°C) within the past 24 hours or significant acute or chronic infection within the previous 7 days
* significant acute or chronic infections requiring systemic antibiotic treatment within the past 14 days
* not available for all the visits scheduled during the study period
* any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives
* participation in another clinical trial within last 90 days or planned for during the study

  * A pregnancy test (urine) on the scheduled day of each vaccination will be required for any female wishing to participate in the study as well as giving basic menstrual cycle information to cover the period in which and individual may be pregnant but this would not be ascertained by the chemical test.

    * Females of childbearing age who have not used or do not plan to use acceptable birth control measures for the duration of the study. Oral, injected or implanted hormonal contraceptive, diaphragm or condom with spermicidal agent or intrauterine device are considered acceptable forms of birth control. If sexually active the subject should have been using one of the accepted birth control methods at least two months prior to study entry.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent and agreement for samples to be sent overseas
* adults and adolescents 16-40 years scheduled to undergo routine tonsillectomy
* in good health at the time of entry into the study as determined by medical history, physical examination and clinical judgment of the investigator
* availability for all the visits scheduled in the study

Exclusion Criteria:

* tonsillectomy for allergic conditions
* receipt of or intent to immunize with any vaccination (other than influenza vaccine or post-exposure tetanus vaccination) or investigational agents within 50 days prior to enrolment and throughout the study period
* previous receipt of any MenB vaccine
* chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs (Inhaled and topical steroids will not be allowed.)
* history of confirmed or suspected meningococcal infection or close contact with an individual with culture or PCR proven N. meningitidis serogroup B within the previous 60 days
* pregnancy (or plans to become pregnant during study)* or breast feeding
* not taking or unwilling to take sufficient measures to avoid pregnancy occurring for the duration of the study period**
* any chronic or progressive disease (eg neoplasm, cardiac, respiratory, liver, gastrointestinal, renal, neurological disease, autoimmune disease, blood dyscrasias or diathesis) or history of dependence/abuse of drugs or alcohol • any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* administration of immunoglobulins and/or any blood products in the last year or planned administration during the study period
* history of any anaphylactic shock, asthma, urticaria or any other allergic reaction after previous vaccinations, or known hypersensitivity to any vaccine component
* fever (oral temperature equal to or greater than 38.5°C) within the past 24 hours or significant acute or chronic infection within the previous 7 days
* significant acute or chronic infections requiring systemic antibiotic treatment within the past 14 days
* not available for all the visits scheduled during the study period
* any condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives
* participation in another clinical trial within last 90 days or planned for during the study * A pregnancy test (urine) on the scheduled day of each vaccination will be required for any female wishing to participate in the study as well as giving basic menstrual cycle information to cover the period in which and individual may be pregnant but this would not be ascertained by the chemical test.

  * Females of childbearing age who have not used or do not plan to use acceptable birth control measures for the duration of the study. Oral, injected or implanted hormonal contraceptive, diaphragm or condom with spermicidal agent or intrauterine device are considered acceptable forms of birth control. If sexually active the subject should have been using one of the accepted birth control methods at least two months prior to study entry.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2009-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
T-cell proliferation following vaccination and its regulation. | After 2 or 3 doses of vaccine

SECONDARY OUTCOMES:
Serum bactericidal antibody and OMV ELISA antibody. | After each does of vaccine
Salivary antibody | After each dose of vaccine
B-cell memory | After 2 or 3 doses of vaccine

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - UBHT, Bristol, Avon
  - North Bristol NHS Trust, Bristol, Avon